CLINICAL TRIAL: NCT07021170
Title: A Double-Blinded Randomized Controlled Trial Comparing Elan Specialized Bariatric Supplements With Standard Multivitamins in Patients Undergoing Sleeve Gastrectomy, Roux-en-Y Gastric Bypass, and One-Anastomosis Gastric Bypass
Brief Title: Trial Comparing Elan Specialized Bariatric Supplements With Standard Multivitamins in Patients Undergoing Bariatric Procedures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Professor of General surgery, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Elan vs Standard Multivitamins
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Vitamin Deficiencies
Keywords: Elan Specialized Bariatric Supplements; Standard Multivitamins; Sleeve Gastrectomy; Roux-en-Y Gastric Bypass; One-Anastomosis Gastric Bypass
MeSH Terms: conditions — Avitaminosis

STUDY DESIGN:
Intervention Model Description: Participants enrolled in the trial will receive one of two oral multivitamin regimens for a total duration of 12 months, commencing on postoperative day 30. Within each surgical subgroup, including SG, RYGB, and OAGB, participants will be randomized in a 1:1 ratio to receive either a specialized bariatric supplement or a standard over-the-counter multivitamin.
  The specialized supplements, developed by Elan, include Elan Believe, Elan Compass, and Elan Supreme. Elan Believe is formulated specifically for patients undergoing SG, Elan Compass is tailored for RYGB and Elan Supreme, designed for OAGB. These zinc levels are aligned with ASMBS recommendations for SG and RYGB and slightly exceed the IFSO guideline of 30 mg/day for OAGB.
  The comparator supplement is a commercially available, over-the-counter multivitamin containing 100% of the recommended daily allowance (RDA) for essential vitamins and minerals.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Elan in Patients Undergoing Sleeve Gastrectomy (Active Comparator): Patients undergoing sleeve gastrectomy and administrating Elan Specialized Bariatric Supplements (Elan Believe)
  Interventions: Dietary Supplement: Elan Believe
- Standard Multivitamins in Patients Undergoing Sleeve Gastrectomy (Active Comparator): Patients undergoing sleeve gastrectomy and administrating Standard Multivitamins (over-the-counter multivitamin containing 100% of the recommended daily allowance (RDA) for essential vitamins and minerals)
  Interventions: Dietary Supplement: Standard Multivitamins
- Elan in Patients Undergoing Roux-en-Y Gastric Bypass (Active Comparator): Patients undergoing Roux-en-Y Gastric Bypass and administrating Elan Specialized Bariatric Supplements (Elan Compass)
  Interventions: Dietary Supplement: Elan Compass
- Standard Multivitamins in Patients Undergoing Roux-en-Y Gastric Bypass (Active Comparator): Patients undergoing Roux-en-Y Gastric Bypass and administrating Standard Multivitamins (over-the-counter multivitamin containing 100% of the recommended daily allowance (RDA) for essential vitamins and minerals)
  Interventions: Dietary Supplement: Standard Multivitamins
- Elan in Patients Undergoing One-Anastomosis Gastric Bypass (Active Comparator): Patients undergoing One-Anastomosis Gastric Bypass and administrating Elan Specialized Bariatric Supplements (Elan Supreme)
  Interventions: Dietary Supplement: Elan Supreme
- Standard Multivitamins in Patients Undergoing One-Anastomosis Gastric Bypass (Active Comparator): Patients undergoing One-Anastomosis Gastric Bypass and administrating Standard Multivitamins (over-the-counter multivitamin containing 100% of the recommended daily allowance (RDA) for essential vitamins and minerals)
  Interventions: Dietary Supplement: Standard Multivitamins

INTERVENTIONS:
Dietary Supplement: Elan Believe — Elan Believe is formulated specifically for patients undergoing SG and contains 18 mg of elemental zinc.
  Arms: Elan in Patients Undergoing Sleeve Gastrectomy
Dietary Supplement: Elan Compass — Elan Compass is tailored for RYGB and contains 24 mg of zinc.
  Arms: Elan in Patients Undergoing Roux-en-Y Gastric Bypass
Dietary Supplement: Elan Supreme — Designed for OAGB, provides 36 mg of zinc.
  Arms: Elan in Patients Undergoing One-Anastomosis Gastric Bypass
Dietary Supplement: Standard Multivitamins — Over-the-counter multivitamin containing 100% of the recommended daily allowance (RDA) for essential vitamins and minerals. Unlike the specialized formulations, the standard multivitamin is not designed to accommodate the altered gastrointestinal absorption characteristics of post-MBS patients.
  Arms: Standard Multivitamins in Patients Undergoing One-Anastomosis Gastric Bypass; Standard Multivitamins in Patients Undergoing Roux-en-Y Gastric Bypass; Standard Multivitamins in Patients Undergoing Sleeve Gastrectomy

SUMMARY:
Obesity has escalated to pandemic levels, impacting over 650 million adults globally and significantly contributing to the burden of non-communicable diseases such as type 2 diabetes, cardiovascular disease, obstructive sleep apnea, non-alcoholic fatty liver disease, and infertility. The chronic, multifactorial nature of obesity presents substantial challenges for long-term management, as lifestyle modifications and pharmacotherapy often yield limited and transient success. In this context, Metabolic and bariatric surgery (MBS) has emerged as the most effective and enduring treatment for obesity, offering significant weight loss and marked improvement or remission of obesity-related comorbidities.

The most prevalent MBS procedures include sleeve gastrectomy (SG), Roux-en-Y gastric bypass (RYGB), and one-anastomosis gastric bypass (OAGB). While these interventions offer considerable metabolic advantages, they inherently cause significant modifications to gastrointestinal anatomy and physiology, which can predispose patients to long-term micronutrient deficiencies. These deficiencies can stem from reduced dietary intake, altered gastric acid secretion, decreased intrinsic factor production, and the bypassing of critical absorptive sites in the gastrointestinal tract. Commonly affected nutrients encompass iron, vitamin B12, Vitamin B6, folate, vitamin D, calcium, and zinc. If not effectively managed, these nutrient deficiencies can lead to anemia, secondary hyperparathyroidism, osteopenia, neurological complications, immune dysfunction, and impaired postoperative recovery.

Population-based recommended dietary allowances (RDAs) and tolerable upper intake levels (ULs) tend to underestimate the nutritional requirements for postoperative patients, as they are derived from healthy cohorts. Many standard formulations may fall short due to inadequate dosages, non-bioavailable forms, or poor tolerability, which can significantly impact patient adherence to supplementation regimens. Over-the-counter multivitamins, such as Centrum®, are designed for the general population and often lack the dosing, bioavailability, or elemental forms required for post-MBS physiology, particularly following bypass procedures.

The American Society for Metabolic and Bariatric Surgery (ASMBS) recommends 8-22 mg of elemental zinc per day, depending on the procedure, and the International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO) and the World Gastroenterology Organization (WGO) recommend up to 30 mg/day for OAGB patients. These values are below the national upper limit in Egypt, which is 25 mg/day.

Moreover, there is evidence indicating a discrepancy in nutrient deficiencies among different bariatric surgery patients; for instance, OAGB patients exhibit a greater prevalence of iron and zinc deficiencies compared to those undergoing RYGB or SG, thereby necessitating proportionally higher supplementation tailored to their specific needs.

DETAILED DESCRIPTION:
Consequently, specialized supplements containing adjusted doses of iron, zinc, and copper, within or slightly exceeding international guideline recommendations, are proposed to address the heightened risk of deficiencies, particularly in MBS procedures such as RYGB and OAGB, which are both clinically necessary and scientifically supported. In response to these shortcomings, specialized MBS supplements have been formulated to meet the unique physiological requirements and anatomical changes associated with each surgical procedure. The Elan Bariatric Supplement line, featuring Elan Believe for sleeve gastrectomy, Elan Compass for Roux-en-Y gastric bypass, and Elan Supreme for omega-loop gastric bypass, illustrates this tailored approach. It combines procedure-specific formulations aimed at optimizing nutrient absorption, minimizing gastrointestinal side effects, and enhancing patient compliance.

Despite the theoretical benefits of these specialized formulations, robust evidence supporting their clinical superiority over standard multivitamins remains scarce. Randomized controlled trials are warranted to ascertain whether these tailored supplements lead to improved nutritional status, enhanced tolerability, and superior overall outcomes in the post-MBS population. The present study intends to bridge this gap by evaluating the incidence of micronutrient deficiencies, along with biochemical and clinical outcomes, and patient compliance over 12 months between individuals receiving specialized Elan supplements and those utilizing standard multivitamins following SG, RYGB, and OAGB. This trial will stratify its analysis based on the type of surgery to assess the differential impacts of supplementation per the distinct anatomical and absorptive characteristics of these three procedures.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants must be adults:

* Aged 18 to 65 years
* Capable of providing informed consent
* Willing to comply with study procedures and follow-up visits over 12 months.
* Candidates must have no prior history of MBS or gastrointestinal surgery and must be scheduled for one of the three aforementioned primary procedures.
* Both male and female patients will be considered, and no restrictions will be placed based on ethnicity or socioeconomic status.

Exclusion Criteria:

Exclusion criteria include:

* The presence of chronic conditions that may independently affect micronutrient metabolism or absorption, such as chronic kidney disease, inflammatory bowel disease, or hepatic insufficiency.
* Additional exclusion criteria include pregnancy or lactation at the time of enrollment
* Plans for pregnancy within the study period
* Active malignancy
* Any use of investigational drugs or supplements within the past 30 days.
* Patients undergoing revisional bariatric surgery or conversion procedures will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 624 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative micronutrient deficiencies at 3, 6, and 12 months following surgery. | 3, 6, and 12 months following surgery.
  Deficiencies will be assessed for six key micronutrients commonly affected by bariatric procedures: iron, vitamin B12, folate, vitamin D, calcium, and zinc. Thresholds for biochemical deficiency will be defined according to institutionally accepted reference ranges and international clinical guidelines. All measurements will be performed on fasting blood samples collected during scheduled follow-up visits.

SECONDARY OUTCOMES:
Measures of compliance | At 6 and 12 months
  Will be assessed using a complementary method: monthly pill counts.
Measures of tolerability | At 3, 6, and 12 months following surgery
  Tolerability will be assessed through systematic reporting of adverse events, with particular attention to gastrointestinal symptoms that may impair adherence. Events will be recorded at each follow-up visit and classified according to severity and their potential relationship to the study supplement.
Changes in biochemical markers (hemoglobin, ferritin, parathyroid hormone, and magnesium) | Over the 12-month follow-up period.
  Biochemical outcomes will also include trends in hemoglobin, ferritin, parathyroid hormone (PTH), and magnesium levels over the 12-month follow-up period.
Anthropometric changes | from enrollment till the end of the study (12 months)
  Changes in BMI (weight and height will be combined to report BMI in kg/m^2) at 3, 6, and 12 months. (weight in kilograms, height in meters)
Anthropometric changes | from enrollment till the end of the study (12 months)
  Changes in body weight and adiposity measure including %EWL (weight in kilograms) at 3, 6, and 12 months. %EWL is defined as the percentage of above-ideal body weight lost.
Compliance with supplementation | Administered at 6 and 12 months
  Compliance with supplementation will be assessed using a complementary method: Validated five-item Medication Adherence Report Scale (MARS-5), administered at 6 and 12 months. The MARS-5 instrument evaluates common non-adherence patterns and yields a cumulative score ranging from 5 to 25, with higher scores indicating greater adherence. Participants will be categorized into three adherence levels: high (scores of 23 to 25), moderate (scores of 20 to 22), and low (scores below 20). These adherence classifications will be used to explore associations between adherence and clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The analysis will be performed on a blinded dataset after completing the medical/scientific review. All protocol violations will be identified and resolved, and the dataset will be declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com), handled according to Good Clinical Practice guidelines, Data Protection Directive certificate, and complied with Title 21 CFR Part 11. Furthermore, the data centers where all the research data will be stored are certified according to ISO27001, ISO9001, and Dutch NEN7510.
  Can be asked by the contact person
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Whole study period
Access Criteria: Ask contact person